CLINICAL TRIAL: NCT00107055
Title: REN-1654 in Sciatica: A Phase 2, Randomized, Double-Blind, Placebo Controlled, Multi-Center Study in Subjects With Pain Due to Lumbosacral Radiculopathy
Brief Title: Study of REN-1654 in Patients With Sciatica Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renovis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: REN-1654-2-03
Record Dates: First submitted 2005-04-04; First posted 2005-04-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Sciatica; Herniated Disc; Radiculopathy
Keywords: Herniated nucleus pulposus; Lumbosacral radiculopathy; Anti-TNF alpha; Tumor necrosis factor alpha
MeSH Terms: conditions — Sciatica; Intervertebral Disc Displacement; Radiculopathy

INTERVENTIONS:
Drug: REN-1654

SUMMARY:
The purpose of this study is to gain initial safety and efficacy data on the experimental agent REN-1654 in patients with pain that radiates down the leg(s), and is typical of sciatica (lumbosacral radiculopathy). These patients will usually have a herniated disc that is causing compression on the nerves coming out of the spinal column.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study to determine the efficacy and tolerability of REN-1654 in subjects with sciatica. After screening and baseline clinical assessments, subjects will be randomly assigned to receive REN 1654 100 mg or matching placebo, once daily for 3 weeks. Leg pain, back pain and other efficacy measures will be assessed at 1 and 3 weeks after initiation of treatment. A subset of patients will undergo analysis of blood levels of REN-1654 during the course of the study (pharmacokinetics). Subjects will discontinue treatment after 3 weeks and return after a further 3 weeks off therapy for a final clinical assessment 6 weeks after initiation of treatment. If a subject does not return for follow-up, an effort will be made by telephone to document their clinical status and whether other interventions have been made.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18 to 55, able and willing to provide written informed consent to participate in the study.
* Able to read, understand and follow the study instructions, including completion of pain intensity rating scales.
* Leg pain radiating to or below the knee in a dermatomal pattern, diagnosed as being due to sciatica or lumbar or lumbosacral radiculopathy, the onset of which occurred 2 to 12 weeks prior to initiation of study treatment.
* Leg pain severity on a screening Categorical Pain Intensity Rating (for the prior 24 hour period) of at least 4, using an 11-point categorical pain intensity scale with 0 = no pain and 10 = worst pain imaginable.
* Leg pain on a screening Categorical Pain Intensity Rating rated as more severe than back pain.
* Positive straight leg raising (SLR) test as defined in Appendix B of this protocol.
* Subjects who are compliant in maintaining a Pain Diary between screening and baseline visits, and who record a 24-hour average Categorical Pain Intensity Rating score of at least 4 or greater on at least 3 days during the week prior to baseline visit.
* Subject who can maintain stable pharmacologic treatments for sciatica symptoms taken prior to dosing including analgesics, anti-inflammatory medications (e.g. NSAIDS), antidepressants, anticonvulsants, anxiolytics, or muscle relaxants. Subjects must be on stable doses of such medications for 2 weeks prior to the baseline visit, and maintained on the same doses throughout the study. Medications taken on an as-needed basis are permitted, and subjects will be asked to record daily usage of such medications in the subject diary.
* Subjects who at screening are receiving adjunctive analgesic therapy such as acupuncture or biofeedback should either discontinue it or establish a schedule of treatments that will remain consistent for 2 weeks prior to the baseline visit, and throughout the study.
* Subject with screening laboratory values within normal limits, or if abnormal must be considered not clinically significant and in the opinion of the Investigator not to place the subjects at risk.
* If female, must be post-menopausal, surgically sterile, not currently pregnant (verified by a screening pregnancy test) or nursing, and using a reliable contraception method such as intrauterine device (IUD), hormonal birth control pills, or double barrier method (male condom, female condom or diaphragm with spermicidal jelly).
* If male, must agree to use double-barrier methods of contraception.

Exclusion Criteria:

* History of peripheral neuropathy or any other pain conditions with pain intensity equal to or greater than the pain associated with sciatica.
* Motor loss in a muscle corresponding to the affected dermatome graded as more than "trace".
* History of cauda equina syndrome, symptomatic scoliosis, spondylolisthesis (degenerative or isthmic), ankylosing spondylitis, rheumatoid arthritis or other inflammatory arthropathies. Degenerative arthritis is allowed.
* History of hepatic, cardiovascular, renal, gastrointestinal, hematological, neurological, endocrine (including diabetes), metabolic, pulmonary, immunological (including HIV infection) or psychiatric disease that in the opinion of the Investigator would pose a significant safety risk for a subject exposed to an investigational compound such as REN-1654.
* History of the following ophthalmic disorders based upon general medical review at the screening visit. Subjects will further undergo a screening ophthalmologic assessment. Should any of the following be identified at the screening ophthalmologic examination, the subject will be excluded from the study.

  * Symptomatic cataract, resulting in any visual impairment (if a subject has been diagnosed with cataract to a degree that the cataract interferes with daily living and/or regarding which an ophthalmologist has recommended cataract surgery);
  * Other vision-impairing disorders (if a subject is aware of any eye disorder that has impaired vision, such as age-related macular degeneration, lazy eye (amblyopia), double vision, or any optic nerve inflammation; presbyopia and other non-pathological visual acuity deficits are not exclusionary);
  * Glaucoma or history of ocular hypertension (intraocular pressures greater than 21 mmHg).
* Cognitive or psychiatric disorders that may diminish compliance with study procedures, including maintenance of a daily pain diary and accurate dosing of study medication.
* Subjects who, at time of enrollment, have requested for or been advised by their physicians to receive local, regional, or spinal (articular, epidural, intrathecal or nerve root block) injections of medications for pain treatment or surgical intervention for their sciatica symptoms.
* Although subjects who report work-related injuries will be allowed to enroll, subjects will be excluded if they are involved in litigation related to the current episode of sciatica.
* Subjects with a screening creatinine laboratory value of ≥ 2.0 mg/dL.
* Screening liver enzyme results greater than the upper limit of the normal range
* Use of chemotherapy agents or history of cancer, other than basal cell carcinoma and squamous cell carcinoma, within five years prior to the screening visit.
* History of drug or alcohol abuse within one year prior to screening.
* Use within 2 weeks before start of study investigational compound dosing at baseline and through the end of the study of any investigational compound, any epidural, intrathecal, or nerve root block agent, corticosteroids, etanercept or other anti-TNF-α agent, topical anesthetics, or topical analgesics .
* Previous participation in another REN-1654 study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2003-12; Study Completion 2005-04

PRIMARY OUTCOMES:
Leg Pain: Change in Average Daily 11-Point Categorical Pain Intensity Rating at the end of the 3-week treatment period

SECONDARY OUTCOMES:
Initiation of the following clinical interventions and time to intervention, if elected, through the 3-week treatment period and 3-week post treatment follow-up period:
[1] Local, regional, or spinal (articular, epidural, intrathecal, or nerve root block) injections of medications for pain treatment. [2] Surgery for treatment of sciatica symptoms
Use of concomitant analgesic medications (tracked by daily log of medication usage)
Back Pain: Change in Average Daily Categorical Pain Intensity
Leg Pain: Change in Maximum (or movement-induced) Daily Categorical Pain Intensity Rating
Back Pain: Change in Maximum (or movement-induced) Daily Categorical Pain Intensity
Change in Oswestry Low Back Disability Questionnaire; Change in Straight Leg Raising test
Change in muscle weakness
Change in sensory deficit
Change in tendon reflexes
Global impression of change: subject and investigator

CONTACTS AND LOCATIONS:
Overall Officials: Randall W Moreadith, MD, PhD, Study Director — Chief Medical Officer, Renovis, Inc.
Locations (19):
- United States (19):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Advanced Clinical Therapeutics, LLC, Tuscon, Arizona
  - Orthopaedic Spine Center at Stanford University Medical Center, Stanford, California
  - Mile High Research Center, Denver, Colorado
  - Clinical Research of West Florida, Clearwater, Florida
  - Renstar Medical Research, Inc., Ocala, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia
  - Brigham & Women's Hospital, Pain Trials Center, Boston, Massachusetts
  - Washington University School of Medicine, Pain Management Center, St Louis, Missouri
  - A&A Pain Institute of St. Louis, St Louis, Missouri
  - Research Across America, New York, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - The Cleveland Clinic Spine Institute, Cleveland, Ohio
  - Lehigh Valley Hospital Neurosciences and Pain Research, Allentown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Central Texas Spine Institute, Austin, Texas
  - Advanced Clinical Research, West Jordan, Utah

REFERENCES:
- [Background] Sommer C, Schafers M, Marziniak M, Toyka KV. Etanercept reduces hyperalgesia in experimental painful neuropathy. J Peripher Nerv Syst. 2001 Jun;6(2):67-72. doi: 10.1046/j.1529-8027.2001.01010.x. PMID 11446385
- [Background] Karppinen J, Korhonen T, Malmivaara A, Paimela L, Kyllonen E, Lindgren KA, Rantanen P, Tervonen O, Niinimaki J, Seitsalo S, Hurri H. Tumor necrosis factor-alpha monoclonal antibody, infliximab, used to manage severe sciatica. Spine (Phila Pa 1976). 2003 Apr 15;28(8):750-3; discussion 753-4. PMID 12698115